CLINICAL TRIAL: NCT04814758
Title: Diffusion-weighted Images as an Additional Method for Diagnosing Histological Types of Nephroblastoma in Children
Brief Title: DWI in the Diagnosis of Histological Types of Nephroblastoma in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCPHOI-2019-08
Record Dates: First submitted 2021-03-04; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-02

CONDITIONS: Nephroblastoma (Wilms Tumour)
Keywords: paediatric; oncology; kidney; DWI; MRI; nephroblastoma; Wilms tumour; quantitative estimation
MeSH Terms: conditions — Wilms Tumor; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MRI DWI sequence (ADC values) — Initially and after pre-operative chemotherapy To evaluate the differences in ADC values according to the malignancy degree of nephroblastoma in children

SUMMARY:
Initially, or after preoperative chemotherapy, patients with a kidney tumor are examined on 3T MR scanner or 1.5T MR scanner. A standard MRI study of the abdomen with contrast enhancement is performed. DWI (diffusion weighted) images are included in the standard investigation package and consist of diffusion maps. Then, using Philips workstation (ISP 9.0, Philips, Netherlands), DWI mapping and ADC values collection (mm2/s) are performed. The placement of region of interest (ROI) is selected in the kidney mass in a solid and cystic area with a size up to 100 mm2.

After the preoperative abdomen MRI, a surgical treatment is performed. Histological material is directed to the pathologist, who carried out the histological staging by the malignancy degree (low, intermediate, high). The data is entered into the database and the relationship between ADC values and histological degrees of malignancy of nephroblastoma is investigated

DETAILED DESCRIPTION:
Initially, or after preoperative chemotherapy, patients with a kidney tumor are examined on 3T MR scanner or 1.5T MR scanner, using 8-channel body coil. A standard MRI study of the abdomen with contrast enhancement is performed. DWI (diffusion weighted) images are included in the standard investigation package and consist of diffusion maps (DWI 3b) with 3 b-factors (50; 600; 800 or others, optional). Then, using Philips workstation (ISP 9.0, Philips, Netherlands), DWI mapping and ADC values collection (mm2/s) are performed. The placement of region of interest (ROI) is selected in the kidney mass in a solid and cystic area with a size up to 100 mm2. The values are entered in the table due to the stage of the chemotherapy.

After the preoperative abdomen MRI, a surgical treatment is performed. Histological material is directed to the pathologist, who carried out the histological staging by the malignancy degree (low, intermediate, high). The data is entered into the database and the relationship between ADC values and histological degrees of malignancy of nephroblastoma is investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Age under 18 y.o.;
2. Renal mass with confirmed histology.

Exclusion Criteria:

1. Absolute contraindications to magnetic resonance imaging (pacemaker, ferromagnetic implants, etc.);
2. Refusal to sign the informed consent.

Ages: 6 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 230 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2023-12-21 (Estimated); Study Completion 2023-12-21 (Estimated)

PRIMARY OUTCOMES:
To evaluate the differences in ADC values according to the malignancy degree of nephroblastoma in children | Point 1. 15 ± 3 days Before the start of therapy - the starting point.
To evaluate the differences in ADC values according to the malignancy degree of nephroblastoma in children | Point 2. after pre-operative chemotherapy up to 1 week

SECONDARY OUTCOMES:
To evaluate the reproducibility and compatibility of the ADC values measurement; | Point 1. 15 ± 3 days Before the start of therapy - the starting point.
To evaluate the reproducibility and compatibility of the ADC values measurement; | Point 2. after pre-operative chemotherapy up to 1 week
To assess the sensitivity and specificity of the MRI DWI sequence (ADC values) in the diagnosis of the malignancy degrees of nephroblastomas in children; | Point 1. 15 ± 3 days Before the start of therapy - the starting point.
To assess the sensitivity and specificity of the MRI DWI sequence (ADC values) in the diagnosis of the malignancy degrees of nephroblastomas in children; | Point 2. after pre-operative chemotherapy up to 1 week
To estimate the differences in ADC values within the intermediate degree of nephroblastoma malignancy in children | Point 1. 15 ± 3 days Before the start of therapy - the starting point.
To estimate the differences in ADC values within the intermediate degree of nephroblastoma malignancy in children | Point 2. after pre-operative chemotherapy up to 1 week
To assess the ADC values change in depending according to the provided chemotherapy. | Point 1. 15 ± 3 days Before the start of therapy - the starting point.
To assess the ADC values change in depending according to the provided chemotherapy. | Point 2. after pre-operative chemotherapy up to 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Galina f Tereshchenko, PhD, Study Director — Chief radiology department at Dmitry Rogachev National Medical Research Center Of Pediatric Hematology, Oncology and Immunology
Locations (1):
- Dmitry Rogachev National Medical Research Centre of Pediatric Hematology, Oncology and Immunology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No